CLINICAL TRIAL: NCT06392724
Title: A Single-arm, Open-label, Single-center Study to Evaluate the Safety and Tolerability of Intravenous GEN6050X Gene Therapy in Ambulatory Boys With Duchenne Muscular Dystrophy (DMD).
Brief Title: A Study to Evaluate the Safety and Tolerability of GEN6050X in Duchenne Muscular Dystrophy.
Acronym: GEN6050XIIT
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Yi Dai, Chief Physician, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GATx-01-IIT-CLINC
Record Dates: First submitted 2024-04-26; First posted 2024-04-30 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2024-07

CONDITIONS: Duchenne Muscular Dystrophy (DMD)
Keywords: Duchenne Muscular Dystrophy; DMD; Gene therapy; Gene editing; Muscular dystrophies; Hereditary neuromuscular disorders
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Muscular Dystrophies

STUDY DESIGN:
Intervention Model Description: Single-arm unblinded, single-center study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- GEN6050X (Experimental): * A single IV infusion of GEN6050X at a dose of 5×10^13 vector genome(VG)/kg body weight
  * Interventions:
    * Genetic: GEN6050X
  Interventions: Genetic: GEN6050X intravenous injection

INTERVENTIONS:
Genetic: GEN6050X intravenous injection — GEN6050X is an intravenously administered human DMD exon 50 skipping base editing drug.

SUMMARY:
The study will evaluate the safety and tolerability of GEN6050X gene therapy in Duchenne muscular dystrophy (DMD) patients amenable to exon 50 skipping.

DETAILED DESCRIPTION:
GEN6050X is an intravenously administered human DMD exon 50 skipping base editing drug containing dual single-stranded adeno-associated virus serotype 9 (ss.AAV9) vectors.

The study is a first-in-human, single-arm, open-label, single-center clinical trial to evaluate safety and tolerability of a single intravenous infusion of GEN6050X in ambulatory boys with DMD. Other objectives include pharmacokinetics, pharmacodynamics, and the preliminary clinical efficacy of GEN6050X over 52 weeks. A total of three ambulatory pediatric participants (aged 4 to 9 years old) are expected to enroll, each receiving a dose of 5×10^13 vg/kg. These participants will be dosed in a staggered fashion.

Safety assessments will include monitoring of adverse events (AEs), laboratory tests, electrocardiograms (ECGs), vital signs, and physical examinations throughout the study duration. In addition, a comprehensive short-term prophylactic immunosuppression regimen(including rituximab and sirolimus) will be administered prior to treatment in order to mitigate potential immune response.

ELIGIBILITY:
Inclusion Criteria:

1. Subject age: 4-10 years old (including 10 years old)
2. Gender: Male
3. Patients with DMD gene exon deletion types confirmed by molecular diagnosis: 8-49, 20-49, 22-49, 51, 51-53, 51-55, 51-57, 51-59, 51-60, 51-67, 51-69, 51-75 or 51-78 and other mutations amenable to exon 50 skipping.
4. The participant is able to walk independently and completes the 10-meter walk test without assistance.
5. Participant is able to complete time to stand from supine independently in less than 30s.
6. The participant is able to cooperate with motor assessment testing.
7. Receipt of glucocorticoids for 6 months and a stable daily dose for at least 12 weeks prior to study entry
8. Ability to tolerate muscle biopsies under anesthesia with no contraindications to these procedures.

Exclusion Criteria:

1. Participants are in the active period of viral infection, including infections such as TORCH virus, Epstein-Barr(EB) virus, and severe acute respiratory syndrome coronavirus 2 (SARS-COV-2).
2. Received a live attenuated vaccine within 3 months prior to receiving GEN6050X, or was exposed to an influenza (or other inactivated) vaccine within 30 days prior to receiving GEN6050X, or received systemic antiviral, anti-infective, and/or interferon therapy.
3. Serological tests found HIV, Hepatitis B Virus(HBV), hepatitis C virus(HCV), and syphilis infection.
4. Severe infection (e.g., pneumonia, pyelonephritis, or meningitis) within 4 weeks prior to receiving gene therapy.
5. With clear symptoms of cardiomyopathy, echocardiography shows that the left ventricular ejection fraction is less than 40%.
6. Need for continuous or intermittent assisted support from a ventilator.
7. Diagnosed with autoimmune disease or receiving related treatment for autoimmune disease.
8. The following indicators are abnormal in laboratory biochemical testing:

   γ-glutamyl transpeptidase (GGT) above the 2-fold upper limit and total bilirubin above 1.5 times the upper limit, cystatin C (cystatin C) > 1.27 mg/L, hemoglobin (Hgb) < 100 or >200 g/L; Leukocytes (WBC) > 18.5×10^9/L or platelet ≤ 125×10^9/L.
9. The titer of AAV9 neutralizing antibody determined by cell suppression assay > 1:50.
10. Patients have received any gene therapy (e.g., adeno associated virus(AAV) gene therapy), cell therapy (e.g., stem cell transplantation), in vivo editing, or ex vivo editing therapy (e.g., CRISPR-Cas9, TALEN) in the past.
11. Participant has any contraindication to immunosuppressive therapy.
12. Has a medical condition or extenuating circumstance that, in the opinion of the principal investigator, is unsuitable for participation in the clinical trial.
13. The family does not wish to disclose the patient's study participation to the attending physician and other medical providers.

Ages: 4 Years to 10 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Estimated)
Dates: Start 2024-07-05 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of GEN6050X measured by incidence of adverse events (AEs). | through 1 year post-treatment
  Incidence of dose-limiting safety or intolerability, as measured by treatment-related adverse events according to Common Terminology Criteria for Adverse Events (CTCAE) V5.0.

SECONDARY OUTCOMES:
Physical Therapy Assessment North Star Ambulatory Assessment (NSAA） | Screening, 6 months-3 Years
  The NSAA measures the quality of ambulation in young boys with Duchenne Muscular Dystrophy.
Physical Therapy Assessment Time to run/walk 10 meters(TTRW) | Screening, 6 months-3 Years
  Change in Time to Run/Walk 10 Meters Test (TTRW)
Physical Therapy Assessment 6MWT | Screening, 6 months-3 Years
  Change in Six-minutes Walk Test (6MWT)
Physical Therapy Assessments Change in Time to Stand (TTSTAND) | Screening, 6 months-3 Years
  Change in Time to Stand (TTSTAND)
Physical Therapy Assessments Ascend and Descend of 4 steps | Screening, 6 months-3 Years
  Change in Time to Climb 4 Steps Test
Physical Therapy Assessments Hand-held dynamometer | Screening, 6 months-3 Years
  The force generated for each muscle strength (elbow extension, elbow flexion, knee extension, and knee flexion on the dominant side only) will be measured by Hand-held dynamometer.
Physical Therapy Assessments upper limb function | Screening, 6 months-3 Years
  Change score in Performance of Upper Limb (PUL) 2.0
Physical Therapy Assessments Pulmonary function | Screening, 6 months-3 Years
  Change in pulmonary function test
Dystrophin protein expression | 24 weeks post-treatment
  Dystrophin protein recovery level in muscle biopsy.
Serum creatine kinase(CK) | through 1 year post-treatment
  Decrease in CK levels in circulating blood

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yuan J, Ma Y, Huang T, Chen Y, Peng Y, Li B, Li J, Zhang Y, Song B, Sun X, Ding Q, Song Y, Chang X. Genetic Modulation of RNA Splicing with a CRISPR-Guided Cytidine Deaminase. Mol Cell. 2018 Oct 18;72(2):380-394.e7. doi: 10.1016/j.molcel.2018.09.002. Epub 2018 Oct 4. PMID 30293782
- See also: Yuan J. et al. Genetic Modulation of RNA Splicing with a CRISPR-Guided Cytidine Deaminase. Mol Cell. 2018 Oct 18;72(2):380-394.e7. — https://pubmed.ncbi.nlm.nih.gov/30293782/